CLINICAL TRIAL: NCT05931536
Title: The Relationship Between Diet, Cognition, Stress, and the Gut Microbiota: A Cross-sectional Study in Healthy Adults
Brief Title: The Relationship Between Diet, Cognition, Stress, and the Gut Microbiota
Acronym: NMB
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Other Study IDs: APC150a
Record Dates: First submitted 2023-06-12; First posted 2023-07-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Microbiota-gut-brain axis; Diet; Cognition; Stress; Dietary fibre
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, saliva, urine, and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low fibre consumers: Healthy adults consuming less than or equal to 18 grams of fibre per day.
  Interventions: Other: Dietary fibre
- Moderate fibre consumers: Healthy adults consuming between 18.1-24.9 grams of fibre per day.
  Interventions: Other: Dietary fibre
- High fibre consumers: Healthy adults consuming greater than or equal to 25 grams of fibre per day.
  Interventions: Other: Dietary fibre

INTERVENTIONS:
Other: Dietary fibre — Habitual dietary consumption from a variety of foods will be assessed using 7-day food logs entered by the participant and assessed for accuracy by a dietitian.

SUMMARY:
This study aims to investigate the relationship between diet and the microbiota-gut-brain axis.

DETAILED DESCRIPTION:
Dietary fibre is well-known for its many health benefits, including the support of gastrointestinal, metabolic, and mental health. Although studies investigating whole dietary patterns in relation to cognition have demonstrated that diet quality and a healthy dietary pattern are associated with better cognitive performance, the role of dietary fibre in this regard is understudied. It is now understood that the gut microbiota (trillions of microbes inhabiting the gastrointestinal tract) communicates bidirectionally with the brain to influence mental health and cognition. Importantly, dietary fibre has been shown to positively affect the microbiota composition. The aim of this study is to understand the effects of dietary fibre on the microbiota-gut-brain axis.

Using a cross-sectional design, habitual low fibre (<=18 grams/day, n=200), moderate fibre (18.1-24.9 grams/day, n=75), and high fibre (=>25 g/day, n=75) consumers will be compared at baseline on measures of cognition, responses to acute and chronic stress, and biological markers of the microbiota-gut-brain axis.

The investigators hypothesize that participants with higher dietary fibre intake at baseline will perform better in the cognitive tasks compared to individuals with low fibre intake, and that this difference can, in part, be mediated by the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be between 18 and 50 years of age.
* Have a body mass index (BMI) between 18.5-29.9 Kg/m2.
* Be in generally good health as determined by the investigator.

Exclusion Criteria:

* Are less than 18 and greater than 50 years of age.
* Have a BMI below 18.5 or above 29.9 Kg/m2.
* Have a significant acute or chronic coexisting illness [cardiovascular, gastrointestinal (GI) [to include functional GI disorders, inflammatory bowel disease, coeliac disease, lactose intolerance, food allergies], immunological, psychiatric [to include formal or as determined by MINI Psychiatric interview, diagnosis of current major depression, anxiety disorder, bipolar spectrum disorder, schizophrenia, other DSM-IV Axis I disorder], neurodevelopmental disorders, immunological, metabolic disorders [to include type I or II diabetes], or any condition which contraindicates, in the investigators judgement, entry to the study.
* Have a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results; all psychoactive medications [to include anxiolytics, antipsychotics, antidepressants, anticonvulsants, centrally acting corticosteroids, and opioid pain relievers), laxatives, enemas, antibiotics, anti-coagulants, over-the counter non-steroidal anti-inflammatories (NSAIDS). Subjects should have a wash-out period of 4 weeks.
* Current prebiotic or probiotic supplement use (a wash-out period of 4 weeks after cessation will allow entry to the study).
* Females who are peri-menopausal, menopausal or post-menopausal.
* Females who are pregnant or planning a pregnancy, or lactating.
* Participants who are not fluent in English.
* Are colour blind.
* Have dyslexia or dyscalculia.
* Are a current habitual daily smoker.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
* Subjects receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Have a malignant disease or any concomitant end-stage organ disease.
* Have completed a study in our laboratory in the past 4 years.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Healthy adult volunteers consuming varying amounts of dietary fibre.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Trait stress/mood: self-report | Compared at baseline
  Self-report questionnaires
Trait stress/mood: hypothalamic-pituitary-adrenal axis activity | Compared at baseline
  Cortisol from saliva samples
Responses to acute stress: self-report | Compared at baseline
  Self-report questionnaires
Responses to acute stress: hypothalamic-pituitary-adrenal axis activity | Compared at baseline
  Cortisol from saliva samples
Responses to acute stress: sympathetic-adrenal-medullary pathway activity | Compared at baseline
  Galvanic skin response taken from the skin on the hand

SECONDARY OUTCOMES:
Cognitive performance: working memory | Compared at baseline
  Spatial Working Memory
Cognitive performance: episodic memory | Compared at baseline
  Modified Rey Auditory Verbal Learning Test (ModRey)
Cognitive performance: decision making | Compared at baseline
  Iowa Gambling Task
Cognitive performance: emotional inhibition | Compared at baseline
  Emotional stroop
Cognitive performance: sustained attention | Compared at baseline
  Rapid Visual Information Processing
Cognitive performance: visual pattern recognition memory | Compared at baseline
  Pattern Recognition Memory
Cognitive performance: cognitive flexibility | Compared at baseline
  Intra-Extra Dimensional Set Shifting
Cognitive performance: social cognition | Compared at baseline
  Emotion Recognition Task
Cognitive performance: affective perceptual bias | Compared at baseline
  Emotional Bias Task
Microbiota composition and function | Compared at baseline
  Shotgun metagenomics of fecal samples
Microbial and host metabolites | Compared at baseline
  Untargeted metabolomics analysis in fecal and urine samples
Inflammation | Compared at baseline
  Inflammatory markers in lipopolysaccharide stimulated and unstimulated bloods

CONTACTS AND LOCATIONS:
Overall Officials: John F Cryan, PhD, Principal Investigator — APC Microbiome Irealnd
Locations (1):
- APC Microbiome Ireland, Cork, Ireland